CLINICAL TRIAL: NCT01900366
Title: Pilot Study for Noninvasive Spectroscopic Detection of Adipose Tissue Inflammation in Obesity
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: JAL-0809
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Obesity
Keywords: Obesity; Healthy Volunteers
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Adipose tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese subjects for fat biopsy: 10 patients recruited during fat biopsies for sample collection
  Interventions: Procedure: Fat Biopsy
- Lean controls for fat biopsy: 5 Lean controls will be recruited
  Interventions: Procedure: Fat Biopsy

INTERVENTIONS:
Procedure: Fat Biopsy — Fat biopsy

SUMMARY:
This study will test the potential of two techniques using light properties of adipose tissue to diagnose crown-like structures and inflammation to be compared with pathologic examination of adipose tissue biopsies from ongoing clinical studies.

DETAILED DESCRIPTION:
Adipose tissue (fat) inflammation is emerging as an important harbinger of disease development including Type 2 diabetes, heart disease and potentially cancer. The hallmark feature of adipose tissue inflammation is the crown-like structure, a dying fat cell surrounded by immune cells attempting to clear the damage. Current methods for detecting adipose tissue inflammation rely on invasive procedures such as fat biopsies. We propose developing methods that use the light reflection properties of inflamed adipose tissue as a potential non-invasive method to detect adipose tissue inflammation.

ELIGIBILITY:
Inclusion Criteria:

-Subjects currently enrolled in a current Rockefeller University study who will be undergoing adipose tissue biopsies as part of the study protocol

Exclusion Criteria:

-History of any skin disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteer and obese subjects
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2013-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Classification of adipose tissue as healthy or inflamed by Raman Spectroscopy | 1 day
  Classification of adipose tissue as healthy or inflamed by Raman Spectroscopy

SECONDARY OUTCOMES:
Steady state oxygenation at the site of tissue biopsy by Diffuse Reflectance Spectroscopy | 1 day
  Steady state oxygenation at the site of tissue biopsy by Diffuse Reflectance Spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Jose Aleman, MD PhD, Principal Investigator — Rockefeller Univesrity
Locations (1):
- The Rockefeller University, New York, New York, United States